CLINICAL TRIAL: NCT06220981
Title: The Oslo Acute Reperfusion Stroke Study (OSCAR)
Acronym: OSCAR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Anne Hege Aamodt, Ass. Prof., Oslo University Hospital
Other Study IDs: 2015-17637
Record Dates: First submitted 2024-01-14; First posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Endovascular treatment

SUMMARY:
Prospective registry of clinical and radiological data in acute ischemic stroke patients after endovascular treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Patients with ischemic stroke and cerebral arterial occlusion treated with endovascular revascularization.
* All stroke severities and vascular distributions are eligible.
* Informed written consent signed by the patient, verbal consent from the patient as witnessed by a non-participating health care person or consent by the signature of the patient's family must be provided before inclusion. Patients for whom no informed consent can be obtained will not be included in the study but will be treated according to standard guidelines.

Exclusion criteria:

• Patient not eligible for the study or not available for follow-up assessments (e.g. non- resident).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: acute ischemic stroke patients with proximal cerebral artery occlusion admitted for endovascular treatment.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2017-01-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Scale Score | 3 months
  Modified Rankin Scale Score (mRS), min 0, max 6

SECONDARY OUTCOMES:
National Institute of Health Stroke Scale Score | discharge
  National Institute of Health Stroke Scale Score (NIHSS, min 0, max 42)
Death due to any cause | 3 months
  Mortality
Infarct volume | 1 day
  Infarct volume (ml)
Incidence of symptomatic intracranial hemorrhage | 1 day
  Incidence of symptomatic intracranial hemorrhage (SICH)
Volume of new areas of diffusion restriction | 1 day
  Volume of new areas of diffusion restriction
serious adverse events | 3 months
  serious adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Enriquez BAB, Skattor TH, Laugesen NG, Truelsen T, Lund CG, Nome T, Beyer MK, Skjelland M, Aamodt AH. External validation of clinical risk prediction score for elderly treated with endovascular thrombectomy. J Neurol. 2024 Sep;271(9):5838-5845. doi: 10.1007/s00415-024-12535-6. Epub 2024 Jul 2. PMID 38954035